CLINICAL TRIAL: NCT03192618
Title: The Impact on Recurrence Risk of Adjuvant Transarterial Chemoinfusion (TAI) for Patients With Hepatocellular Carcinoma And Microvascular Invasion (MVI) After Hepatectomy : A Random, Controlled, Stage III Clinical Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-006-01
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Procedure: adjuvant transarterial chemoinfusion (TAI); Drug: mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
- control group (No Intervention)

INTERVENTIONS:
Procedure: adjuvant transarterial chemoinfusion (TAI) — transarterial chemoinfusion (TAI) with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
  Arms: treatment group
Drug: mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU) — oxaliplatin, calcium folinate, and 5-FU
  Arms: treatment group

SUMMARY:
To compare The Impact on Recurrence Risk of Adjuvant Transarterial Chemoinfusion (TAI) for Patients With Hepatocellular Carcinoma And Microvascular Invasion (MVI) After Hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 75 years;
* ECOG PS<3;
* proven hepatocellular carcinoma with MVI according pathological examination;
* not previous treated for tumor;
* tumor was removed in operation;
* no recurrence occurence at 4 to 7 weeks after surgery;
* the lab test could meet: neutrophil count≥1.5×109/L; hemoglobin≥80g/L; platelet count≥60×109/L; serum albumin≥28g/L; total bilirubin<3-times upper limit of normal; ALT<5-times upper limit of normal; AST<5-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 6 seconds; INR≤2.3;
* sign up consent;
* unrolled by other clinical trials about hepatocellular carcinoma.

Exclusion Criteria:

* cannot tolerate TAI;
* CNS or bone metastasis exits;
* known history of other malignancy;
* be allergic to related drugs;
* underwent organ transplantation before;
* be treated before (interferon included);
* known history of HIV infection;
* known history of drug or alcohol abuse;
* have GI hemorreage or cardiac/brain vascular events within 30 days;
* pregnancy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From date of randomization until the date of recurrence, assessed up to 60 months
  disease-free survival

SECONDARY OUTCOMES:
recurrence rate | 1 year, 2 year, 3 year, 5 year after surgery
  recurrence rate
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun Yat-Sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li SH, Mei J, Cheng Y, Li Q, Wang QX, Fang CK, Lei QC, Huang HK, Cao MR, Luo R, Deng JD, Jiang YC, Zhao RC, Lu LH, Zou JW, Deng M, Lin WP, Guan RG, Wen YH, Li JB, Zheng L, Guo ZX, Ling YH, Chen HW, Zhong C, Wei W, Guo RP. Postoperative Adjuvant Hepatic Arterial Infusion Chemotherapy With FOLFOX in Hepatocellular Carcinoma With Microvascular Invasion: A Multicenter, Phase III, Randomized Study. J Clin Oncol. 2023 Apr 1;41(10):1898-1908. doi: 10.1200/JCO.22.01142. Epub 2022 Dec 16. PMID 36525610
- [Derived] Li S, Mei J, Wang Q, Guo Z, Lu L, Ling Y, Xu L, Chen M, Zheng L, Lin W, Zou J, Wen Y, Wei W, Guo R. Postoperative Adjuvant Transarterial Infusion Chemotherapy with FOLFOX Could Improve Outcomes of Hepatocellular Carcinoma Patients with Microvascular Invasion: A Preliminary Report of a Phase III, Randomized Controlled Clinical Trial. Ann Surg Oncol. 2020 Dec;27(13):5183-5190. doi: 10.1245/s10434-020-08601-8. Epub 2020 May 16. PMID 32418078